CLINICAL TRIAL: NCT05974319
Title: The Effect of Dry Heat and Dry Cold Application on Pain, Anxiety and Fear Levels Before Blood Sample Collection in School Age Children: A Randomized Controlled Study
Brief Title: The Effect of Dry Heat and Dry Cold Application on Blood Sampling in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berna Eren Fidancı, Associate professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GHF_MC1
Record Dates: First submitted 2023-07-11; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: School Age Children; Blood; Procedural Pain; Procedural Anxiety; Fear
Keywords: Blood sampling; Children; Dry heat; Dry cold; Pediatric nurse
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Before blood sampling, the participants were assigned to the experiment 1-dry heat application, experiment 2-dry cold application and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): During the blood sample collection, the application was carried out in line with the routine care.
- Dry heat application (Experimental): The region where the invasive intervention will be performed will be determined by the nurse in charge of the shift. The researcher will heat the thermoregulated electric pad and set it to 42°C. After making sure that there are no contraindications in the application of the electric pad device, a dry heat of 42°C will be applied to the determined area with the electric pad for 5 minutes.
  Interventions: Other: Dry heat application
- Dry cold application (Experimental): The region where the invasive intervention will be performed will be determined by the nurse in charge of the shift. After the researcher is sure that there are no contraindications in the application of the gel pad, dry cold will be applied to the determined area with the gel pad for 3 minutes.
  Interventions: Other: Dry cold application

INTERVENTIONS:
Other: Dry heat application — Dry heat application: The region where the invasive intervention will be performed will be determined by the nurse in charge of the shift. The researcher will heat the thermoregulated electric pad and set it to 42°C. After making sure that there are no contraindications in the application of the electric pad device, a dry heat of 42°C will be applied to the determined area with the electric pad for 5 minutes.
  Arms: Dry heat application
Other: Dry cold application — Dry cold applicaiton: The region where the invasive intervention will be performed will be determined by the nurse in charge of the shift. After the researcher is sure that there are no contraindications in the application of the gel pad, dry cold will be applied to the determined area with the gel pad for 3 minutes.
  Arms: Dry cold application

SUMMARY:
The study was conducted as a parallel group randomized controlled in order to determine the effects of dry heat and dry cold application before blood collection in school-aged children (7-12 years old) on pain, anxiety and fear levels.

Participants were randomly assigned to experiment 1-dry hot application group, experiment 2-dry cold application group and control group.

In Experiment 1-Dry Heat Application group, a dry heat of 42°C was applied to the determined area with an electrical heating pad for 5 minutes before blood sample was taken.

In Experiment 2-Dry Cold Application group, dry cold was applied to the area determined with a gel pad for 3 minutes before blood sample was taken.

In the Control group, blood sampling was performed according to the clinical routine, and no heat or cold application was made.

DETAILED DESCRIPTION:
Prior to blood sampling, parents and children were initially informed about the study in Experiment 1-dry heat, Experiment 2-dry cold, and control groups, and their written and verbal consents were obtained. After obtaining consent, information about the child and family was collected by the researcher with the "Child-Family Introductory Information Form" before the procedure. After the family and the child were introduced to the measurement tools (Wong Baker Faces Pain Scale, Child Fair Anxiety Scale and Medical Procedures Fear Inventory) to be scored, it was explained to the child that his mother or father would be with him during the procedure, and he was taken to the intervention room. Before the blood sample collection, the child's fear and anxiety were evaluated using Child Fear Anxiety Scale.

In Experiment 1-Dry Heat Application group, the electrical heating pad with temperature regulation was heated by the researcher and set to 42°C. After making sure that there were no contraindications (deterioration of skin integrity, etc.) in the application of the electrical heating pad device, a dry heat of 42°C was applied to the determined area with an electrical heating pad for 5 minutes.

In Experiment 2-Dry Cold Application group, dry cold was applied to the determined area with a gel pad for 3 minutes after the researcher made sure that there were no contraindications (deterioration of skin integrity, etc.) in the application of the gel pad.

In the Control group, blood sampling was performed according to the clinical routine, and no heat or cold application was made.

ELIGIBILITY:
Inclusion Criteria:

* 7-12 years old
* Absence of physical and mental illness
* Absence of auditory, visual and verbal speech disability
* Parents' willingness to participate in the research, and signing the volunteer form

Exclusion Criteria:

* Those who do not meet the inclusion criteria
* Those who do not volunteer to participate

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Wong Baker Faces Pain Rating Scale | One minutes after blood sampling; once
  Refers to the pain felt due to the blood sample collection process.

SECONDARY OUTCOMES:
Child Fear Scale | Two minutes before blood sampling, Two minutes after blood sampling; twice.
  It expresses the fear of taking a blood sample, which is a painful procedure.
Child Anxiety Scale | Two minutes before blood sampling, two minutes after blood sampling; twice.
  It expresses the anxiety of taking a blood sample, which is a painful procedure.
Medical Procedures Fear Inventory | Three minutes after blood sampling; once.
  It refers to evaluating children's fears towards medical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Eren Fidancı, RA, Study Director — University of Sağlık Bilimleri
Locations (1):
- Sağlık Bilimleri University Gulhane Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

REFERENCES:
- [Derived] Cil M, Fidanci BE. The effect of dry heat and dry cold application on pain, anxiety and fear levels before blood sample collection in school age children (7-12 years): A randomized controlled study. J Pediatr Nurs. 2023 Nov-Dec;73:e401-e408. doi: 10.1016/j.pedn.2023.10.008. Epub 2023 Oct 19. PMID 37863785